CLINICAL TRIAL: NCT02531997
Title: A Mind-body Intervention to Improve Body and/or Self Image: a Phase II Randomized Trial
Brief Title: A Mind-body Intervention to Improve Body and/or Self Image
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Breast Cancer Research Foundation (Other)
Responsible Party: Principal Investigator, Debra L. Barton, Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HUM00100709
Record Dates: First submitted 2015-08-19; First posted 2015-08-25 (Estimated); Last update posted 2017-12-12 (Actual); Status verified 2017-12

CONDITIONS: Breast Cancer; Ovarian Cancer; Uterine Cancer; Cervical Cancer
Keywords: self-image; sexual health; breast cancer; gynecologic cancer; ovarian cancer; cervical cancer; uterine cancer; mind body; hypnotic relaxation therapy; hypnosis; progressive muscle relaxation
MeSH Terms: conditions — Breast Neoplasms; Ovarian Neoplasms; Uterine Neoplasms; Uterine Cervical Neoplasms | interventions — Autogenic Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hypnotic Relaxation Therapy (Active Comparator): Hypnotic relaxation will be performed in three sessions, two weeks apart, over 6 weeks. The hypnosis sessions will build on each other in terms of content.
  Interventions: Behavioral: Hypnotic Relaxation Therapy
- Progressive Muscle Relaxation (PMR) (Other): The PMR will consist of progressive tensing and relaxing of the muscles from head to toe to a soothing sound of the participant's choosing.
  Interventions: Behavioral: Progressive Muscle Relaxation

INTERVENTIONS:
Behavioral: Hypnotic Relaxation Therapy — There are 3 induction scripts that build upon each other, each about 20 minutes in length. The first focuses on relaxation, feelings of wellness, wholeness, strength, and confidence. The second focuses more on body image related to sexuality, sexual desire, passion, and romanticism. The third includes suggestions from the previous inductions, but adds a behavior that the woman chooses to incorporate for the last 2 weeks of the intervention. A digital recording will be provided of the intervention content for home practice.
  Arms: Hypnotic Relaxation Therapy
Behavioral: Progressive Muscle Relaxation — Women will be instructed how to do progressive relaxation and will be given the opportunity to ask questions and express concerns. The research therapist will utilize a script to focus the conversation on relaxation and planning the implementation of the behavior. Participants will be given a digital recording of 4 pleasant background sounds to facilitate their relaxation practice. Home practice will be encouraged.
  Arms: Progressive Muscle Relaxation (PMR)

SUMMARY:
The purpose of this study is to determine if hypnotic relaxation therapy is a more effective intervention for improving self-image in women who have been diagnosed with breast or gynecologic cancer when compared to progressive muscle relaxation therapy.

DETAILED DESCRIPTION:
This will be a phase II randomized controlled trial involving two arms: hypnotic relaxation and progressive muscle relaxation (PMR), using a 2:1 randomization schedule.

1. Evaluate the impact of a hypnotic relaxation intervention compared to progressive muscle relaxation on body image distress.

   Hypothesis 1: Women randomized to the hypnotic relaxation will have significantly more improvement in body image distress as measured by the Impact of Treatment Scale than women randomized to receive progressive muscle relaxation at 6 weeks.
2. Evaluate the impact of a hypnotic relaxation intervention compared to progressive relaxation on sexual self-image, sexual health, and mood.

   Hypothesis 2: Women randomized to hypnotic relaxation will show significantly more improvement on the Sexual Self-Schema Scale, the Patient Reported Outcomes Measurement Information System (PROMIS) sexual health scale and the Positive-Negative Affect Scale (PANAS) than women receiving progressive relaxation at 6 weeks.
3. Evaluate the side effects of hypnotic and progressive muscle relaxation. Hypothesis 3a: Hypnotic relaxation will not be associated with significantly more negative side effects than progressive muscle relaxation.

   Hypothesis 3b: Neither hypnotic nor progressive muscle relaxation will be associated with negative side effects.
4. Explore the physiologic effects of hypnotic relaxation compared to progressive muscle relaxation by evaluating cortisol slopes and comparing am/pm cortisol values.

Hypothesis 4a: Women receiving hypnotic relaxation will have a steeper cortisol slope, higher am and lower pm cortisol concentrations at the end of 6 weeks compared with women receiving progressive muscle relaxation.

Women will be referred from providers in the Breast and Gynecology Clinics of the University of Michigan Cancer Center as well as the Symptom Management, Sexual Health and Psycho-Oncology clinics. The study coordinator will provide education about the trial and a consent form will be provided for review. If a woman decides to participate, she will sign the consent form. Sessions will be held at Dr. Barton's behavioral research office located on Washtenaw Avenue in Ann Arbor, where there is privacy, a recliner, a relaxing environment, and convenient parking.

Both intervention arms will involve three sessions that will occur at 2 week intervals. Each visit will last about 40 minutes to an hour.

ELIGIBILITY:
Inclusion Criteria:

* a history of any stage of breast or gynecologic cancer
* reported a change in body/self-image since diagnosis and wish to improve it. Two screening questions will be used: Has body image or self-image changed in an unwanted way since the cancer diagnosis? (Answer must be yes.) Would the potential participant like to be able to do something to improve body image or self-image? (Answer must be yes.)
* Concurrent cancer treatment of any kind is allowed, but the participant can also have completed all treatment
* Performance status of 2 or better

Exclusion Criteria:

* Diagnosis of a major depressive episode, an acute anxiety disorder, psychosis, or schizophrenia as listed in the patient's medical history per Diagnostic and Statistical Manual for Mental Health-IV criteria in the chart and/or by self-report
* Past history of sexual abuse.
* Currently on 2 or more antidepressant therapies for mood disturbance of any kind. Past use is allowed, just not current use.
* Currently on 2 or more anti-anxiety therapies. Past use is allowed, just not current use.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Impact of Treatment Scale | Change from baseline at 6 weeks
  This scale is a measure of body change stress and was developed by investigators at The Ohio State University. It was developed and tested specifically in women with breast cancer and then edited a little and tested in women with gynecologic cancer. It has demonstrated good reliability and validity in both samples, with Cronbach alphas over .90, and was able to discriminate between women with lower and higher satisfaction with their sexual life.

SECONDARY OUTCOMES:
Sexual Self-Schema Scale for Women | Change from baseline at 6 weeks
  This scale was developed by investigators from The Ohio State University (OSU) in female undergraduates at OSU and was later tested in a group of community women and subsequently in women with gynecologic cancer and breast cancer. It is a measure of 26 trait adjectives that are self-rated from 0 (not descriptive of me) to 6 (very much descriptive of me). Three dimensions have been demonstrated: passionate/romantic; open/direct and embarrassed/conservative. Cronbach's alpha has been demonstrated to be .76.
PROMIS Sexual Health Measure | Change from baseline at 6 weeks
  The PROMIS initiative is a large effort supported by the National Institute of Health and was created in such a way that investigators can use items that are relevant to the population and research question while maintaining validity. Most of the measures were developed in the cancer population. The sexual function and satisfaction measure is one tool that has good content, face, discriminant, and convergent validity, and is, therefore, ready to be incorporated into clinical trials. It demonstrates good convergent validity with the Female Sexual Function Index (FSFI), which is considered the gold standard measure in sexual function, but PROMIS is shorter and easier to score. The global satisfaction domain with 7 items (correlation of 0.76 with the FSFI satisfaction subscale) and interest domain with 4 items (correlation of 0.84 with the FSFI desire subscale) with two questions about interfering factors (hot flashes and fatigue) for a total of 13 items are being used.
Positive/Negative Affect Scale (PANAS) | Change from baseline at 6 weeks
  The PANAS was developed as a brief measure to evaluate self-reported mood, focusing on positive and negative affect. Conceptually, positive affect represents a state of high engagement and enthusiasm whereas negative affect represents a state of distress and lack of engagement. It contains 20 items, 10 measuring positive affect and 10 measuring negative affect. It has high internal consistency (.88 PA and .85 NA) when participants answer about their feelings in the past few days. The scale was developed in an undergraduate student population, but since development, it has been used in a wide range of populations including women with breast cancer.
Global Impression of Change, effort and satisfaction | End of study about 6 weeks
  The Subject Global Impression of Change is a 7-point item in which the participant rates the change in the overall status since beginning the study (ranging from "very much better," "moderately better," "a little better," "about the same," "a little worse," "moderately worse," to "very much worse"). It has been used extensively for determination of minimally clinically significant differences in numerous oncology clinical trials. This tool measures perception of benefit from the study intervention by the participant.

OTHER OUTCOMES:
Self-Report Side Effect Questionnaire | Weekly through end of study about 6 weeks
  Using the numeric analog scale of 0 (none) to 10 (as bad as it can be), women will be asked to answer a number of questions about potential negative experiences related to the intervention.
Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 | Weekly for 6 weeks
  This is a provider grading scale used in National Cancer Institute Clinical Trials. The adverse events that will be assessed and graded in this trial based on relevancy are the psychiatric disorders: agitation, anxiety, insomnia, restlessness personality change and psychoses.
Practice Log days | Daily through end of study about 6 weeks
  A daily log that was developed by the investigator to measure days of practice.
Practice Log minutes | Daily through end of study about 6 weeks
  A daily log that was developed by the investigator to measure minutes of practice.

CONTACTS AND LOCATIONS:
Overall Officials: Debra Barton, RN, PhD, FAAN, Principal Investigator — University of Michigan School of Nursing
Locations (1):
- University of Michigan School of Nursing, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
Small pilot study for feasibility and effect size. Data would not be helpful to others; too small for secondary analysis.

REFERENCES:
- [Derived] Arring NM, Lafferty CK, Clark PM, Barton DL. The experience of women in a phase II trial of hypnosis and progressive muscle relaxation for body image: informing future research questions. J Psychosoc Oncol. 2024;42(1):148-158. doi: 10.1080/07347332.2023.2206406. Epub 2023 Apr 28. PMID 37114974